CLINICAL TRIAL: NCT03660501
Title: Continuous Vital Sign Monitoring During Admission for Acute Exacerbations of Chronic Obstructive Pulmonary Disease - an Observational Study
Brief Title: Wireless Assessment of Respiratory and Circulatory Distress in Chronic Obstructive Pulmonary Disease - an Observational Study
Acronym: WARD-COPD
Status: Completed | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Technical University of Denmark (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Mikkel Elvekjaer, MD, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: WARD-COPD_v1.1
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Continuous monitoring
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Troponin, Arterial Blood Gas
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Continuous monitoring system — Patients recruited will be continuously monitored with Isansys Lifetouch patch, Isansys wireless blood pressure monitor, Nonin WristOx 3150, Empatica E4, and Radiometer TCM5 FLEX monitor.

SUMMARY:
For patients admitted to the medical ward, it is often difficult to predict if their clinical condition will deteriorate, however subtle changes in vital signs are usually present 8 to 24 hours before a life-threatening event such as respiratory failure leading to ICU admission, or unanticipated cardiac arrest. Such adverse trends in clinical observations can be missed, misinterpreted or not appreciated as urgent. New continuous and wearable 24/7 clinical vital parameter monitoring systems offer a unique possibility to identify clinical deterioration before patients condition progress beyond the point-of-no-return, where adverse events are inevitable. The WARD-COPD project aims to determine the correlation between cardiopulmonary micro events and clinical adverse events during the first four days after hospital admission with acute exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted with AECOPD
* Recruitment and monitoring start is possible within 24 hours after admission

Exclusion Criteria:

* Patient expected not to cooperate
* Patient allergic to plaster, plastic or silicone
* Active therapy withdrawn
* Patients with dementia or not able to give informed consent
* Patients with pacemaker or implantable cardioverter-defibrillator (ICD) unit
* Expected discharge within less than 24 hours from possible inclusion

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients admitted to hospital with acute exacerbation of COPD will be included in the study upon arrival to the medical ward.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Any serious adverse events | within 30 days after inclusion
  E.g. cardiac arrest, ICU admission, acute myocardial infarction, stroke, sepsis, acute kidney injury or other serious adverse events (defined in Protocol Appendix A)

SECONDARY OUTCOMES:
Mortality | within 6 months after inclusion
Readmission | within 6 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyhoff, MD, PHD, Study Chair — Bispebjerg and Frederiksberg Hospital
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Gentofte Hospital, Hellerup

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elvekjaer M, Rasmussen SM, Gronbaek KK, Porsbjerg CM, Jensen JU, Haahr-Raunkjaer C, Molgaard J, Sogaard M, Sorensen HBD, Aasvang EK, Meyhoff CS. Clinical impact of vital sign abnormalities in patients admitted with acute exacerbation of chronic obstructive pulmonary disease: an observational study using continuous wireless monitoring. Intern Emerg Med. 2022 Sep;17(6):1689-1698. doi: 10.1007/s11739-022-02988-w. Epub 2022 May 20. PMID 35593967